CLINICAL TRIAL: NCT04470648
Title: COVID-19 Infection at Samusocial in Paris: Descriptive and Serological Survey
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Samusocial de Paris (Unknown); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: C20-50
Record Dates: First submitted 2020-07-12; First posted 2020-07-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2023-02

CONDITIONS: SARS-COV2 Infection
Keywords: Seroprevalence; SARS-COV2; Precarious
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood for serology testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hosted in the center and HCWs at the epidemic period: people hosted in the health care or in the women center and health care workers working in one these centers during the epidemic time.
  People with initial positive SARS-COV2 serology will have a second blood test to mesure atibodies kinetic
  Interventions: Diagnostic Test: blood test for SARS-COV2 serology

INTERVENTIONS:
Diagnostic Test: blood test for SARS-COV2 serology — each person who will accept to participate will have a bood test for a SARS-COV2 serology

SUMMARY:
Study of COVID-19 seroprevalence in precarious population living in shelters of Samusocial de Paris and in staff working in these centers during COVID-19 epidemic.

DETAILED DESCRIPTION:
After emergence of a new coronavirus (Severe Acute Respiratory Syndrome Coronavirus 2, SARS-CoV2) responsible for a cluster of respiratory infection at Wuhan, China, on January, 7th 2020, first cases were diagnosed in France in January 24th 2020.

Health care components of Samusocial de Paris (Lits Haltes Soins Santé (LHSS)) were created in 2006. They provide medical care for homeless people and people in social distress not needing an hospitalization. Sometimes there are 3 persons in a bedroom.

In december 2018, a special shelter for isolated women or women in precarious situations opened.

Because of the living conditions in these centers and the difficulty for these populations to respect social distancing and hygiene recommendations.

A first case of COVID-19 was identified on March 8th 2020 in one of these healthcare centers. Other cases were detected in the same center, then in another center on March 16th, then in the dormitory of the women shelter on March 30th.

A recent study showed an important prevalence of SARS-COV2 in residents of a homeless shelter in Boston (36%), most of them were asymptomatic.

Seroprevalence studies are done in general population or in health care workers, but don't include vulnerable people.

It seemed important to us to describe the epidemic in these centers and to study COVID-19 seroprevalence in these particular populations.

ELIGIBILITY:
Inclusion Criteria:

* to have been hosted or working in one the three centers (LHSS Ridder-Plaisance or Saint Michel or Halte femmes) between march and may 2020
* to be aged 18 y or more
* to be able to give an informed consent

Exclusion Criteria:

* people who refuse to participate
* not being able to give an informed consent
* Person subject to a legal protection measure (safeguard of justice, curatorship or guardianship)
* Person who does not understand the information provided on how to carry out the research
* Obstacle to venous sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people hosted and workers at one these 3 centers during the epidemic time (march to may 2020)
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
SARS-COV-2 seroprevalence in 3 centers for homeless and people in social distress | 6 months
  Primary objective is to evaluate SARS-COV2 seroprevalence in people hosted and health care workers of 3 centers of Samusocial de Paris where COVID19 epidemics occured

SECONDARY OUTCOMES:
Morbidity rate | 6 months
  Measure of morbidity in the participating population in the 3 centers
Covid-19 related death rate in the 3 centers from March to May 2020 | 6 months
  Number of deaths related to Covid-19 during the epidemic in the 3 centers
Ratio of negative serology rate and positive serology rate in the 3 centers | 6 months
Ratio of SARS-COV2 seroprevalence obtained in these centers to the estimated seroprevalence in the Ile de France region | 6 months
kinetics of SARS-COV2 antibodies in people with initial positive serology | 10 months
  2 blood tests 4 and 8 months afetr the first one

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan Yazdanpanah, MD PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Haltes pour femmes, Paris
  - LHSS Saint-Michel, Paris
  - LHSS Ridder-Plaisance, Paris

REFERENCES:
- [Background] Bernard Stoecklin S, Rolland P, Silue Y, Mailles A, Campese C, Simondon A, Mechain M, Meurice L, Nguyen M, Bassi C, Yamani E, Behillil S, Ismael S, Nguyen D, Malvy D, Lescure FX, Georges S, Lazarus C, Tabai A, Stempfelet M, Enouf V, Coignard B, Levy-Bruhl D; Investigation team. First cases of coronavirus disease 2019 (COVID-19) in France: surveillance, investigations and control measures, January 2020. Euro Surveill. 2020 Feb;25(6):2000094. doi: 10.2807/1560-7917.ES.2020.25.6.2000094. PMID 32070465
- [Background] Lescure FX, Bouadma L, Nguyen D, Parisey M, Wicky PH, Behillil S, Gaymard A, Bouscambert-Duchamp M, Donati F, Le Hingrat Q, Enouf V, Houhou-Fidouh N, Valette M, Mailles A, Lucet JC, Mentre F, Duval X, Descamps D, Malvy D, Timsit JF, Lina B, van-der-Werf S, Yazdanpanah Y. Clinical and virological data of the first cases of COVID-19 in Europe: a case series. Lancet Infect Dis. 2020 Jun;20(6):697-706. doi: 10.1016/S1473-3099(20)30200-0. Epub 2020 Mar 27. PMID 32224310
- [Background] Deslandes A, Berti V, Tandjaoui-Lambotte Y, Alloui C, Carbonnelle E, Zahar JR, Brichler S, Cohen Y. SARS-CoV-2 was already spreading in France in late December 2019. Int J Antimicrob Agents. 2020 Jun;55(6):106006. doi: 10.1016/j.ijantimicag.2020.106006. Epub 2020 May 3. PMID 32371096
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Backer JA, Klinkenberg D, Wallinga J. Incubation period of 2019 novel coronavirus (2019-nCoV) infections among travellers from Wuhan, China, 20-28 January 2020. Euro Surveill. 2020 Feb;25(5):2000062. doi: 10.2807/1560-7917.ES.2020.25.5.2000062. PMID 32046819
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Baggett TP, Keyes H, Sporn N, Gaeta JM. Prevalence of SARS-CoV-2 Infection in Residents of a Large Homeless Shelter in Boston. JAMA. 2020 Jun 2;323(21):2191-2192. doi: 10.1001/jama.2020.6887. PMID 32338732
- [Result] Husain M, Rachline A, Cousien A, Rolland S, Rouzaud C, Ferre VM, Gomez MV, Le Teurnier M, Wicky-Thisse M, Descamps D, Yazdanpanah Y, Charpentier C, Pasquet-Cadre A. Impact of the COVID-19 pandemic on the homeless: results from a retrospective closed cohort in France (March-May 2020). Clin Microbiol Infect. 2021 Oct;27(10):1520.e1-1520.e5. doi: 10.1016/j.cmi.2021.05.039. Epub 2021 Jun 7. PMID 34111590